CLINICAL TRIAL: NCT00211159
Title: Omega-3 Fatty Acid Treatment of 174 Patients With Mild to Moderate Alzheimer's Disease (OmegAD): a Randomized Double-blind Trial
Brief Title: OmegAD (Omega-3 and Alzheimer's Disease)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: OmegAD#1
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2005-04

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; Omega-3 fatty acid; Dietary supplementation; Cognition; Safety
MeSH Terms: conditions — Alzheimer Disease

INTERVENTIONS:
Drug: EPAX 1050TG

SUMMARY:
Memory loss and difficulties with thinking associated with Alzheimer's disease (AD) may be due to a deficiency in the brain of a fatty acid named DHA. The aim of this trial is to see if dietary supplementation with a preparation, rich in DHA, will halt cognitive impairment in AD patients

ELIGIBILITY:
Inclusion Criteria: Alzheimer's disease with MMSE 15-30, living in own homes, treated with stable dose of acetylcholine esterase inhibitor for >3 months and remaining on that treatment for the study period

Exclusion Criteria: Already treated with omega-3 fatty acids, NSAIDs, warfarin, being an alcohol abuser, suffering from serious concomitant disease or not having a caregiver

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 204
Dates: Start 2000-12

PRIMARY OUTCOMES:
Cognition measured according to ADAS-cog, MMSE scales

SECONDARY OUTCOMES:
Safety, tolerability, blood pressure
Gene expression | 2007-2018
  mRNA expression and DNA methylation changes in blood leukocytes in relation to changes of plasma and cerebrospinal concentrations of omega-3 fatty acids
Dose-response studies in relation to APOE4 status, to body weight and to gender | 2007-2018
  Analysis of changes of plasma and cerebrospinal fluid concentrations of omega-3 fatty acids in relation to APOE4 status, body weight and gender, as well as to changes in ADAS-cog and MMSE as measures of cognition.

CONTACTS AND LOCATIONS:
Overall Officials: Tommy Cederholm, MD, PhD, Principal Investigator — Uppsala University, Sweden
Locations (1):
- Karolinska University Hospital Huddinge, Stockholm, Sweden

REFERENCES:
- [Background] Eriksdotter M, Vedin I, Falahati F, Freund-Levi Y, Hjorth E, Faxen-Irving G, Wahlund LO, Schultzberg M, Basun H, Cederholm T, Palmblad J. Plasma Fatty Acid Profiles in Relation to Cognition and Gender in Alzheimer's Disease Patients During Oral Omega-3 Fatty Acid Supplementation: The OmegAD Study. J Alzheimers Dis. 2015;48(3):805-12. doi: 10.3233/JAD-150102. PMID 26402079
- [Result] Freund-Levi Y, Eriksdotter-Jonhagen M, Cederholm T, Basun H, Faxen-Irving G, Garlind A, Vedin I, Vessby B, Wahlund LO, Palmblad J. Omega-3 fatty acid treatment in 174 patients with mild to moderate Alzheimer disease: OmegAD study: a randomized double-blind trial. Arch Neurol. 2006 Oct;63(10):1402-8. doi: 10.1001/archneur.63.10.1402. PMID 17030655
- [Result] Wang X, Hjorth E, Vedin I, Eriksdotter M, Freund-Levi Y, Wahlund LO, Cederholm T, Palmblad J, Schultzberg M. Effects of n-3 FA supplementation on the release of proresolving lipid mediators by blood mononuclear cells: the OmegAD study. J Lipid Res. 2015 Mar;56(3):674-681. doi: 10.1194/jlr.P055418. Epub 2015 Jan 23. PMID 25616438
- [Result] Freund-Levi Y, Vedin I, Hjorth E, Basun H, Faxen Irving G, Schultzberg M, Eriksdotter M, Palmblad J, Vessby B, Wahlund LO, Cederholm T, Basu S. Effects of supplementation with omega-3 fatty acids on oxidative stress and inflammation in patients with Alzheimer's disease: the OmegAD study. J Alzheimers Dis. 2014;42(3):823-31. doi: 10.3233/JAD-132042. PMID 24934544
- [Result] Freund Levi Y, Vedin I, Cederholm T, Basun H, Faxen Irving G, Eriksdotter M, Hjorth E, Schultzberg M, Vessby B, Wahlund LO, Salem N Jr, Palmblad J. Transfer of omega-3 fatty acids across the blood-brain barrier after dietary supplementation with a docosahexaenoic acid-rich omega-3 fatty acid preparation in patients with Alzheimer's disease: the OmegAD study. J Intern Med. 2014 Apr;275(4):428-36. doi: 10.1111/joim.12166. Epub 2014 Jan 11. PMID 24410954
- [Result] Vedin I, Cederholm T, Freund-Levi Y, Basun H, Garlind A, Irving GF, Eriksdotter-Jonhagen M, Wahlund LO, Dahlman I, Palmblad J. Effects of DHA-rich n-3 fatty acid supplementation on gene expression in blood mononuclear leukocytes: the OmegAD study. PLoS One. 2012;7(4):e35425. doi: 10.1371/journal.pone.0035425. Epub 2012 Apr 24. PMID 22545106
- [Derived] Faxen-Irving G, Falahati F, Basun H, Eriksdotter M, Vedin I, Wahlund LO, Schultzberg M, Hjorth E, Palmblad J, Cederholm T, Freund-Levi Y. Does Fatty Acid Composition in Subcutaneous Adipose Tissue Differ between Patients with Alzheimer's Disease and Cohabiting Proxies? J Alzheimers Dis. 2018;61(2):515-519. doi: 10.3233/JAD-170359. PMID 29154271
- [Derived] Karimi M, Vedin I, Freund Levi Y, Basun H, Faxen Irving G, Eriksdotter M, Wahlund LO, Schultzberg M, Hjorth E, Cederholm T, Palmblad J. DHA-rich n-3 fatty acid supplementation decreases DNA methylation in blood leukocytes: the OmegAD study. Am J Clin Nutr. 2017 Oct;106(4):1157-1165. doi: 10.3945/ajcn.117.155648. Epub 2017 Aug 30. PMID 28855224
- [Derived] Vedin I, Cederholm T, Freund-Levi Y, Basun H, Hjorth E, Irving GF, Eriksdotter-Jonhagen M, Schultzberg M, Wahlund LO, Palmblad J. Reduced prostaglandin F2 alpha release from blood mononuclear leukocytes after oral supplementation of omega3 fatty acids: the OmegAD study. J Lipid Res. 2010 May;51(5):1179-85. doi: 10.1194/jlr.M002667. Epub 2009 Nov 24. PMID 19965584
- [Derived] Vedin I, Cederholm T, Freund Levi Y, Basun H, Garlind A, Faxen Irving G, Jonhagen ME, Vessby B, Wahlund LO, Palmblad J. Effects of docosahexaenoic acid-rich n-3 fatty acid supplementation on cytokine release from blood mononuclear leukocytes: the OmegAD study. Am J Clin Nutr. 2008 Jun;87(6):1616-22. doi: 10.1093/ajcn/87.6.1616. PMID 18541548
- [Derived] Freund-Levi Y, Basun H, Cederholm T, Faxen-Irving G, Garlind A, Grut M, Vedin I, Palmblad J, Wahlund LO, Eriksdotter-Jonhagen M. Omega-3 supplementation in mild to moderate Alzheimer's disease: effects on neuropsychiatric symptoms. Int J Geriatr Psychiatry. 2008 Feb;23(2):161-9. doi: 10.1002/gps.1857. PMID 17582225